CLINICAL TRIAL: NCT05540795
Title: Diagnostic Accuracy of 3T Unenhanced MR Imaging for the Detection of Parathyroid Lesions Before Surgery in Hemodialysis Patients With Secondary Hyperparathyroidism Comparison With 4DCT
Brief Title: Diagnostic Accuracy of 3T MR for Secondary Hyperparathyroidism Comparison With 4DCT
Status: Completed | Type: Observational
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Ying Wang, Director, Fifth Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: ZDWY.HYXK.006
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Parathyroid Gland Disease; Secondary Hyperparathyroidism
MeSH Terms: conditions — Parathyroid Diseases; Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Secondary hyperparathyroidism (SHPT) is a common serious complication in the maintenance process of hemodialysis patients, characterized by diffuse or nodular hyperplasia of parathyroid glands. Parathyroidectomy for patients with drug-refractory SHPT is recommended in the clinical practice guidelines of the Global Organization for Improving Prognosis in Kidney Disease (KDIGO) and the Japanese Dialysis Therapy Society (JSDT) . Therefore, accurate localization and detection of parathyroid abnormalities is the key to avoid persistent recurrence of the disease. However, the sensitivity and specificity of the existing ultrasound and 99MTC-MIBI diagnosis are limited. CT examination is radiative and requires iodine contrast medium with nephrotoxicity, which may require timely dialysis and long-term monitoring for hemodialysis patients. 3T MRI has no radiation and does not need to use iodine contrast agent, which can well detect parathyroid lesions . Previous studies have reported that 3T MRI can diagnose primary hyperparathyroidism (PHPT), but the diagnostic efficacy of SHPT is still unclear. Therefore, this study aims to evaluate the preoperative diagnostic value of non-enhanced 3T MRI compared with 4DCT in patients with secondary hyperparathyroidism after hemodialysis.

DETAILED DESCRIPTION:
MR examinations were performed by using the 3 Tesla unit (Siemens Magnetom Verio, Siemens Medical Solutions) with a dedicated eight-channel neurovascular phased array coil. The field of view was adjusted to include the area from the angle of the mandible to the level of the tracheal carina. The protocol included an axial and a coronal T1-weighted fast spin-echo (FSE) sequence, an axial T2-weighted FSE sequence with Dixon fat saturation, and a coronal and sagittal T2-weighted FSE sequence with inversion recovery fat saturation.

4DCT images were scanned with the 128-section dual-source multi-detector row unit (Somatom Definition Flash; Siemens Medical Solutions). All patients were scanned from the angle of the mandible to the carina. The 4DCT protocol included the acquisition of unenhanced images followed by the acquisition of arterial and delayed (venous) phase image series. Unenhanced images were obtained by using the following parameters: a collimation of 64×0.6 mm, 120 kVp for the deliverance of a dose-modulated amperage of 250 mAs, a pitch of 0.7, and a gantry rotation time of 0.28 seconds. The arterial and venous phase scans was performed in dual-energy mode with a dual source of 80 kVp and 140 kVp tube voltages using the following parameters: tube current-time product 230 and 89 mAs, respectively; collimation, 64 × 0.6 mm; rotation speed, 0.28 seconds; and helical pitch, 0.7. The arterial and venous phase scanning began automatically at 10 s and 35 s after the left common carotid artery reached the trigger attenuation threshold (100 HU) using automated scan-triggering software (CARE Bolus CT; Siemens Healthineers). The volume of iodinated contrast material (iohexol, Omnipaque 300; GE Healthcare, SH, China) was 70 mL, and the injection rate was 3 mL/s. The mean dual-source CT dose index volume was 34.5 mGy.

The sensitivity and specificity as well as the positive-predictive and negative-predictive values (PPV, NPV) of each imaging modality for preoperative parathyroid hyperplasia localization to the correct quadrant were compared. For the per-quadrant localization, if a lesion was suspected to be parathyroid hyperplasia by the imaging report and was correlated with the surgical and pathology results, this was interpreted as a true-positive lesion. Otherwise, if the lesion was not confirmed to be parathyroid hyperplasia during surgery, this was considered to be a false-positive case. If a lesion was not reported by the radiologist in the exact quadrant but was present during surgery and histopathologic examination, this was regarded as a false-negative lesion.

ELIGIBILITY:
Inclusion Criteria:

* 1) undergoing total parathyroidectomy with severe SHPT, and 2) undergoing 4DCT and routine unenhanced MRI.

Exclusion Criteria:

* Patients were excluded if they had known contraindications to MR or CT imaging. Patients were also excluded if their images could not be used for diagnosis due to quality.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with severe SHPT who were receiving maintenance hemodialysis and had undergone parathyroidectomy were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-05-28 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
sensitivity | 1month
  The number of positive tests as a percentage of the total number of cases

CONTACTS AND LOCATIONS:
Overall Officials: Ying Wang, MD, Principal Investigator — Fifth Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- FifthSunYetSen, Zhuhai, Guangzhou, China